CLINICAL TRIAL: NCT05639062
Title: Narrative-based Card Game (NCG) in Improving Spiritual Well-being, Enhancing Hope, Decreasing Psychological Symptoms, and Promoting Quality of Life Among Chinese Childhood Cancer Patients: A Pilot Randomized Controlled Trial
Brief Title: Narrative-based Card Game in Improving Spiritual Well-being Among Chinese Childhood Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCG
Record Dates: First submitted 2022-11-07; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Pediatric Cancer
Keywords: spiritual well-being; intervention; childhood cancer patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative-based card game (Active Comparator)
  Interventions: Behavioral: Narrative-based card game
- PUKE card game (No Intervention)

INTERVENTIONS:
Behavioral: Narrative-based card game — This intervention aims to evaluate the preliminary effects of narrative-based card game intervention on spiritual well-being, hope, anxiety, depressive symptoms, and QoL of childhood cancer patients at postintervention and at 1-, and 3-month follow-up postintervention.
  Arms: Narrative-based card game

SUMMARY:
Cancer as a life-threatening disease can trigger children's unique spiritual needs. Unmet spiritual needs can cause low level of spiritual well-being, which is a central component for the overall quality of life (QoL) of cancer patients and was inversely associated with depressive symptoms, anxiety and a low level of hope. However, there has been no intervention focused on improving spiritual well-being among childhood cancer patients. Evidence from adult cancer patients suggests that narrative intervention can effectively address spiritual needs and improve spiritual well-being, while playing card game can combine an emotionally sensitive topic with an enjoyable activity, providing insight into the development of narrative-based card games for childhood cancer patients. The first objective of this pilot study is to assess the feasibility of narrative-based card game among Chinese childhood cancer patients. The second objective is to evaluate the preliminary effects of narrative-based card game intervention on spiritual well-being, hope, anxiety, depressive symptoms, and QoL of childhood cancer patients at postintervention and at 1-, and 3-month follow-up postintervention.

DETAILED DESCRIPTION:
A pilot randomized controlled trial will be carried out. A convenience sample of 60 children with cancer will be recruited. Subjects who are randomized into the experimental group which will participate the narrative-based card game or into the control group which will play a PUKE card game only for entertainment purpose, that mimics the time and attention of the intervention. Feasibility measures (i.e., the eligibility rate, consent rate, randomization rate etc.) will be collected immediately after the completion of the intervention. Also, all subjects will be asked to complete structured questionnaires to assess their spiritual well-being, hope, anxiety, depressive symptoms, and QoL at postintervention and at 1-, and 3-month follow-up postintervention.

ELIGIBILITY:
Inclusion Criteria: (1) age 12-17 old (2) diagnosed with any type of cancer and currently undergoing active treatment (3) knowing about their cancer diagnosis, and (4) able to communicate with Chinese.

-

Exclusion Criteria: (1) those with identified cognitive and/or behavioural problems which affected their verbal communication; (2) those with advanced cancer, including nonresponsive to treatment, stage IV solid tumor that had recurred or progressed as defined, or physician estimated poor prognosis of <60%.

-

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
The length of recruitment | baseline
  The time used for subject recruitment
Eligibility rate | baseline
  The number of eligible childhood cancer patients divided by the number of childhood cancer patients screened prior to eligibility assessment
Consent rate | baseline
  The number of eligible childhood cancer patients who agree to participate divided by the number of eligible childhood cancer patients
Randomization rate | baseline
  The number of participants who are randomized divided by the number of consenting children
Attendance rate | post-intervention
  The number of participants in the experimental group who complete the intervention divided by the number of participants randomized into the group
Retention rate | post-intervention, and 1-month, 3- month follow ups
  The number of participants who remain in the study divided by the number of participants randomized. Retention rate will be calculated at baseline and follow ups.
Completion rate | post-intervention, and 1-month, 3-month follow ups
  The number of participants who complete the questionnaire divided by the number of questionnaires distributed.
Missing data | post-intervention, 1-month, 3- month follow ups
  The percentage of missing data.
Adverse events | post-intervention, 1-month, 3-month follow ups
  Unfavorable or unintended events during the study period that were not present at baseline or appear to have worsened since baseline.

SECONDARY OUTCOMES:
The Chinese version of adapted Functional Assessment of Chronic Illness Therapy Spiritual Well-being Scale at 3 months follow-up | at 3-months follow-up
  Assessing the spiritual well-being of participants, the score for the Chinese version of adapted Functional Assessment of Chronic Illness Therapy Spiritual Well-being Scale is 0-60, with higher scaores indicating higher spiritual well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Q, Ho KY, Lam KKW, Wong FKY, Lam W, Cheng F, Wei H, Chan K, Ting M, Yang FN, Xiao P, Luo T, Wang HX, Yorke J. Preliminary effectiveness and feasibility of an integrated hope techniques and narrative-based card game intervention for pediatric cancer patients in China: a randomized controlled trial. BMC Med. 2025 Jul 31;23(1):449. doi: 10.1186/s12916-025-04287-5. PMID 40745312